CLINICAL TRIAL: NCT03067155
Title: CMV Specific T Cell Therapy for the Treatment of Relapsing or Therapy Refractory CMV Infection After Allogeneic Stem Cell Transplantation With a CMV-positive Donor.
Brief Title: CMV Specific T Cell Therapy After Allogeneic Stem Cell Transplantation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-TJT1401; 2013-004953-26 (EudraCT Number); BHS-TC13 (Other: Belgian Hematological Society)
Record Dates: First submitted 2016-10-06; First posted 2017-03-01 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Hematological Malignancies; CMV Infection
Keywords: allogeneic stem cell transplantation; CMV reactivation
MeSH Terms: conditions — Hematologic Neoplasms; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): The patients for which a suitable donor product can be obtained will be included in the treatment arm of the protocol. Treatment consists of the administration of CMV-specific T-cells, administered through intravenous transfusion. Depending on response in viral load and GVHD status, a second and/or third administration is possible.
  Interventions: Genetic: CMV-specific T cells
- Control group (Active Comparator): Patients for which the investigator can't obtain a suitable donor product, will be included in the control group consisting of standard anti-viral treatment.
  Interventions: Drug: Standard anti-viral therapy

INTERVENTIONS:
Genetic: CMV-specific T cells
  Arms: Treatment group
Drug: Standard anti-viral therapy — Continue with the anti-viral treatment as per standard of care.
  Arms: Control group

SUMMARY:
Viral infections remain an important cause of morbidity and mortality after allogeneic stem cell transplantation (SCT), especially after myelo-ablative conditioning and if the donor is antigen-mismatched or haplo-identical.. In the described setting the patient's own immune system has been destroyed by the necessary highly immuno- and myelo-ablative conditioning and all memory against infections has been deleted. Therefore, there is a high risk for several viral infections and other infectious organisms.Both primary viral infections and reactivations can occur, and patients can become refractory to antiviral treatments, or in some cases an adequate antiviral treatment is unavailable or too toxic. In this study, the investigators will target CMV, as refractory CMV infection and disease is accompanied by an extremely high mortality rate and therefore the development of new treatment approaches is required. Despite the available antiviral drugs, a considerable number of patients are facing an insufficient control of CMV reactivation after SCT. Because reconstitution of CMV-specific T cells confer protection against the development of CMV disease after SCT, attempts have been made to restore antiviral immunity by direct infusion of CMV-specific T cells. Most clinical cellular immunotherapy protocols for CMV treatment have used CMV-specific cytotoxic CD8+ T-cell lines generated by repetitive in vitro stimulation with CMV antigens with success. Despite the proven efficacy, use of cellular therapy in the clinic has been limited, because the approach is time and labor consuming and requires specialized facility allowing handling of the therapeutic cells according to good manufacturing practice. In addition, no sustained response was seen after adoptive transfer that involved only cytotoxic CD8+ T cells. This phenomenon is supported by the fact that recall responses to latent infections depend on the presence of CD4+ T cells to help cytotoxic CD8+ T cells. An alternative approach for the transfer of T-cell immunity is the isolation of Ag-specific T cells ex vivo from the blood of CMV seropositive donors, based on interferon γ (IFN-γ) secretion of T cells after in vitro stimulation with viral Ag, resulting in a combination of CD4+ T helper and cytotoxic CD8+ CMV specific T cells. Using this strategy, a short-term ex vivo protocol was developed for the isolation of pp65 (CMV immunodominant protein)-specific T cells. Since then, several centers have used this protocol in the clinic, infusing low numbers of pp65-specific T cells, that were able to restore protective T-cell immunity against CMV in a post SCT setting in patients with refractory CMV disease or viremia. For this protocol the investigators have set up and validated this method of CMV-specific T-cell generation in the Ghent University Hospital and the investigators will make it available for other Belgian transplant centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  1. All underlying diseases that form an indication for allogeneic stem cell transplantation
  2. Underwent allogeneic stem cell transplantation with a donor that fulfills the following criteria:
* CMV-seropositive at the time of transplant and
* Age 18-70 years 3) Having a CMV reactivation or primary infection or disease with the following characteristics: CMV PCR at least twice positive AND CMV infection relapsing after 3 successful treatment episodes with gancyclovir OR Refractory to treatment with available antiviral drugs which is defined as follows: Persistent positive CMV PCR > detection limit 14 days after initiation of antiviral treatment OR increasing CMV viral load 7 days after initiation of antiviral treatment 4) Informed consent given
* Donor:

  1. Is identical to donor of the previous stem cell transplant
  2. The donor will be pre-screened for the presence of sufficient numbers of CMV-specific T cells:
* IFNgamma producing T cells upon CMVpp65 stimulation are at least twice the background level (unstimulated cells)
* At least 10 events of IFNgamma positive T cells are measured
* IFNgamma producing T cells upon CMVpp65 stimulation are equal or higher than 0,1% of the viable CD4+ and CD8+ cell population If the donor shows sufficient number of circulating CMV-specific cells, according to the test described in 2 3) Only if the donor shows sufficient number of circulating CMV-specific cells, according to the test described in 2:
* Donor has positive IgG serology for CMV, IgM negative or positive
* Donor has signed informed consent for the donation of donor lymphocyte cells
* Donor is found fit for donation by a medical doctor according to selection criteria conform KB annex II (C-2009/18414)
* Donor is negative for infectious disease markers including HCV, HBV and HIV-NAT testing: HBs antigen, HBc/HBs antibodies, Syphilis (TPHA or equivalent), HVC and HIV antibodies.
* Additional testing should be performed and negative when relevant: malaria, west nile virus, trypanosomiasis, HTLV conform KB annex II (C-2009/18414)
* HCG negative within 7 days of apheresis

Exclusion Criteria:

* Patients:

  1. HIV, HCV, HBV positive (HbSAg positivity after vaccination is allowed)
  2. Life expectancy severely limited by disease other than malignancy or viral infection
  3. Administration of cytotoxic agent(s) for cytoreduction within three weeks prior to initiation of the treatment or to be expected within 8 weeks after administration of the treatment
  4. Terminal organ failure except for renal failure (dialysis acceptable)
  5. Uncontrolled other infection than the one being treated
  6. Karnofsky performance score < 60%
  7. Patient is a fertile man or woman who is unwilling to use contraceptive techniques during and for 12 months following treatment
  8. Patient is a female who is pregnant or breastfeeding
  9. Patient with active aGVHD grade 3 or more
  10. Patient with severe chronic GVHD
  11. Patient on corticosteroids > 0.5mg/kg. Patient can still be on therapeutic doses of immunosuppressive therapy, but these will be tapered to the lowest possible dose, as is part of standard care in case of CMV reactivation.
  12. Patient that has received ATG < 1 month prior to infusion or Campath < 1 year prior to infusion
  13. Any condition not fulfilling inclusion criteria
* Donor:

  1. Any condition not fulfilling inclusion criteria

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for whom the investigator can manufacture a product that meets release criteria, and can therefore receive the product. | Within 1 year after the last follow-up visit of the last patient.
  Starting from patients and donors that fulfill all inclusion criteria and do not have any exclusion criterium, and donors fulfilling all pre-apheresis criteria.
Safety of the administered cell product in terms of Graft-versus-Host-Disease occurence/worsening. | Within 1 year after the last follow-up visit of the last patient.
  Evaluation of the frequency of patients who develop de novo or recurrent (with a history of (completely recovered)) acute GVHD grade 2 or more or show worsening of an existing aGVHD with at least 1 grade, or emergence of an additional organ involved.

SECONDARY OUTCOMES:
Clinical efficacy measured by change in CMV PCR or resolution of CMV disease. | Within 1 year after the last follow-up visit of the last patient.
  Clinical efficacy has already been shown (albeit not in a randomized phase 3 trial) but as there is no alternative therapy for these patients (except for continuing the therapy they are already getting and to which they are not (longer) responding, this study is not placebo or best supportive care controlled, but is designed as a single arm study. However, by including all patients who can get the product in the treatment arm and those who can't get the product in the observational arm, the study will be able to have a control group without randomization.
Evaluation of infusion related adverse event as per CTCAE 4.03. | Within 1 year after the last follow-up visit of the last patient.
Explore the relationship between the presence of CMV specific T cells in the peripheral blood of the patient and the objective clinical response | Within 1 year after the last follow-up visit of the last patient.
Make the treatment of relapsing or refractory CMV infection after allogeneic stem cell transplantation with CMV-specific T cell therapy from the CMV positive donor available for patients in Belgium | Within 1 year after the last follow-up visit of the last patient.
Compare resistance to antiviral therapy in both arms (investigational vs. observational) b measuring change in CMV PCR or evaluating resolution of CMV disease. | Within 1 year after the last follow-up visit of the last patient.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Kerre, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (8):
- Belgium (8):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - ZNA Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Université de Liège, Liège
  - Heilig Hart Ziekenhuis Roeselare, Roeselare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geurten C, Ghinai R, Munford H, Lawson S. Efficacy of Cytomegalovirus Specific Immunoglobulins to Reduce CMV Reactivation in Pediatric Hematopoietic Stem Cell Transplant Recipients. J Pediatr Hematol Oncol. 2023 Jan 1;45(1):e82-e86. doi: 10.1097/MPH.0000000000002553. Epub 2022 Sep 22. PMID 36162011